CLINICAL TRIAL: NCT05247151
Title: The Association of Affective Resonance With Empathy Modulated by Negative Symptomatology and Oxytocin
Acronym: OXY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Kerem Böge, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3000194
Record Dates: First submitted 2021-11-08; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Schizophrenia Spectrum Disorders
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Active Comparator): The patients received either a spray of the synthetic oxytocin (24 I.U. Syntocinon®) with mindfulness-bases grow therapy (MBGT) as a positive social context in each condition. Due to an effect latency of 30-80 mins after intranasal administration of oxytocin on social behavior, the dose was administered 30 min before the 50-min session.
  Interventions: Other: Oxytocin
- Placebo (Placebo Comparator): The patients received either a spray of the synthetic placebo (24 I.U.) with mindfulness-bases grow therapy (MBGT) as a positive social context in each condition. Due to an effect latency of 30-80 mins after intranasal administration of oxytocin on social behavior, the dose was administered 30 min before the 50-min session.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Oxytocin — Oxytocin nasal spray in a positive social setting.
  Arms: Oxytocin
Other: Placebo — Placebo nasal spray in a positive social setting.
  Arms: Placebo

SUMMARY:
In previous studies the neuropeptide oxytocin has been in particular associated with social enhancing and anxiety relieving effects.

The purpose of this study is to investigate the effect of oxytocin on empathy in patients with schizophrenia. On a neurobiological level, social effects mediated by oxytocin are based on oxytocin's influence on the complexly regulated mesocorticolimbic dopamine system. Preliminary studies have already shown that oxytocin increases neuronal connections between social reward expectancy networks and networks for socioemotional processes in the brain, which on a behavioral level leads to increased social activation, motivation, and also improved social perception. Furthermore, an increase in empathy modulated by the amygdala has been shown in healthy individuals following oxytocin administration. In particular, primary psychotic disorders, such as schizophrenia, are associated with deficits in the domain of social cognition, including empathy, with the degree of negative symptoms playing an important mediating role. Another study demonstrated a significantly lower expression of empathy as well as a significantly lower oxytocin level in patients with schizophrenia compared to healthy subjects. According to the hypothesis of social salience, which describes an increased importance of certain social stimuli, the effect of oxytocin varies depending on specific contexts and individual variables of the perceiving person, such as the degree of negative symptoms. Therefore, based on such preliminary findings, the research project will explore an effect of oxytocin on empathy within a positively experienced and controlled context, especially in patients with schizophrenia regarding their negative symptoms.

DETAILED DESCRIPTION:
The study design is based on an experimental, double-blinded (participants, instructor), placebo-controlled, proof-of-concept randomized, trial and complies with the CONSORT guidelines. The study was approved by the ethical committee of the Charité - Universitätsmedizin Berlin (EA4/196/19). All study-relevant measures were based on the current Declaration of Helsinki. After eligibility screening, informed consent was obtained at least 24 hours before participants started baseline assessments. Participants were randomly allocated to the experimental condition with admission of oxytocin or to a placebo treatment as the active control condition with MBGT as a positive social context in each condition. Randomization was performed by an independent researcher using a random computer-generated sequence with randomly permuted block sizes. To exclude gender bias, both men and women were included in mixed-gender groups on a balanced basis.

On two dates within one week the application of oxytocin (OXT) nasal spray or placebo took place by trained physicians to test a possible influence of OXT on empathy and other variables in dependence of and the pre-existing expression of a negative symptomatology and a positive social context in form of two psychologically supervised manual-based mindfulness based group sessions (MBGT). Empathy as primary outcome as well as negative symptoms as secondary outcome, and exploratory affect, stress and mindfulness were measured using validated self- and external-rated psychometric questionnaires. Secondary outcomes were conducted merely for exploratory reasons. All outcomes, including venous-blood sampling for OXT plasma levels, were measured before the first session at baseline (T0), after completion of the treatment period of 1-week (T3) and in between after the first session (T1) and before 2nd session (T2). For their time, participants received a financial compensation of 30 Euros after completion of post-intervention assessment.

The patients received either a spray of the synthetic oxytocin (24 I.U. Syntocinon®) or a commercially available nasal spray placebo. P: According to the manufacturer, the nasal sprays for OXT (Syntocinon) and placebo were not distinguishable by appearance, taste, or different rates of ADRs. The choice of dose is based on preliminary studies of optimal effects on aspects of social cognition. Due to an effect latency of 30-80 mins after intranasal administration of OXT on social behavior, the dose was administered 30 min before the 50-min session. The bottles of the nasal sprays were numbered to guarantee blinding of the participants and the treatment team. By applying OXT exclusively before the controlled exercise setting and the refraining from a continuous administration of OXT for one week, reinforcement of negative experiences according to the OXT salience hypothesis outside the created context of the exercises should be avoided. Oxytocin, which is also produced as an endogenous hormone, acts in the human body at Oxytocin receptors in various organ systems. Oxytocin nasal spray (Syntocinon) is used to promote milk let-down in women, who have difficulty breastfeeding and in secondary hypogalactia.

As a positive social context during the placebo-controlled oxytocin application participants attended two supervised MBGT sessions (50 mins each) in groups of 3-6 individuals for a period of one week.

MBGT depicts a novel and innovative treatment program for SSD which was specifically developed within an iterative and participatory research design by our research group MBGT was selected as a positive social context because of explicit feedback from prior studies of participants with schizophrenia spectrum disorders (SSD) that they had felt comfortable during the relevant sessions. Overall, the sessions are taking into account original recommendations for implementing mindfulness in psychosis as well as patient feedback.

Within the sessions, short periods of meditation are used to avoid prolonged periods of silence, and basic anchoring techniques and easily comprehensive language were used according to recommendations.

The two sessions of the manual, which were considered most appropriate with regard to a positive social setting for individuals with SSD, were tailored to the relevant requirements in the context of this study. They focused on two of four core aspects of mindfulness (breath and senses in nature) while interacting with other participants, sharing experiences and expressing emotions, as well as engaging in activities together and enhancing mutual understanding and trust.

The sessions followed a standardized but adapted procedure described in the manual.

They started with an introduction to the topic of the session (breathing or senses in nature), after which 15 mins of mindfulness exercises were practiced based on the topic. Lastly, there were 10 min of sharing experiences, based on the inquiry model as well as 5 min for sharing individual aims.

The first session "Mindfulness of breathing" focused on making participants aware of their own breathing within the present moment and introducing the concept of mindfulness. After an introduction phase within the group, basic psychoeducation about mindfulness and two breathing exercises followed. In form of an inquiry process, participants were able to share their experiences and thoughts with the group.

In the session "Mindfulness of the senses in nature" participants started with a self-reflection phase about the meaning of mindfulness in their every-day life, which they could share with the group. This was followed by an exercise, activating all senses within the present moment and a mindful walk through the nature. After each participant's option to share their experiences with the group, the session was finished with a final resumé by each participant.

The sessions were led by a psychotherapist with over ten years of experience in mindfulness-based practices together with a psychotherapist in training in cognitive behavioral therapy with over three years of experience in mindfulness practice. The sessions were implemented outside within a naturalistic setting due to the restrictions of the hospital in the context of the Covid-19 pandemic and the resulting ban on conducting outpatient groups indoors.

The manual-based sessions are established procedures in each case, for which no risks have been found to have occurred so far on the basis of diverse preliminary work. Adverse effects on participants were notexpected. It nonetheless was ensured by regular feedback from the participants.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Psychiatric diagnosis from the schizophrenic spectrum (ICD-10: F2x.x spectrum) for group of patients
* Mild to moderate positive symptoms (5 < positive symptoms on individual items using P-PANSS)
* Age: 18 - 65 years
* German should either be the mother tongue or spoken at a native level.

Exclusion Criteria:

* Acute psychotic episode with severe positive symptoms (ICD-10: F2 spectrum, 5 ≥ positive symptoms on individual items using P-PANSS).
* Acute suicidality
* Acute consumption phase of a substance dependence, except nicotine
* No severe physical impairments, neurological diseases and e.g. severe craniocerebral trauma e.g. early childhood brain damage

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Change in empathy | Change from baseline (before intervention) to directly after intervention.
  Measured via the Interpersonal Reactivity Index (SPF-IRI). The IRI assesses four dimensions of empathic responding (Perspective taking, Empathic concern, Personal distress, Fantasy) on a 5-point Likert scale ranging from "Does not describe me well" (1) to "Describes me very well" (5). Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Change of negative symptoms | Change from baseline (before intervention) to directly after intervention.
  Measured via the Self-Evaluation of Negative Symptoms (SNS) scale. It is a 20-item self-reported questionnaire with five subscales, namely Alogia, Avolition, Anhedonia, Social withdrawal and Diminished emotional range. Participants can estimate the answer to each question on a scale from 0 (strongly disagree) to 2 (strongly agree). Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Zierhut, Dr., Principal Investigator — Charitè - Universitätsmedizin Berlin; Eric Hahn, PD, Study Director — Charitè - Universitätsmedizin Berlin
Locations (1):
- Charité Universitätsmedizin Berlin, Campus Benjamin Franklin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No